CLINICAL TRIAL: NCT07060937
Title: Clinimetric Properties of Performance Based Functional Outcome Measure After Coronary Artery Bypass Graft (CABG) Surgery
Brief Title: Clinimetric Properties of Performance Based Functional Outcome Measure After (CABG) Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Zarish Ayub
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; CABG
Keywords: Clinimetric properties; Performance based functional outcomes; Time up and go test; Five times sit to stand test; 2 minute walk test; 6 minute walk test
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post CABG surgery patients (Experimental): The intervention includes 30-50 years old male and female post-CABG surgery patients. They will be recruited according to the inclusion criteria of the study and all baseline measurements will be taken from each participant to ensure readiness for the tests performed. The participants will undergo functionality based performance tests which include 5 Time sit to stand test, Time up and go test, 2 Minute walk test and 6 Minute walk test on post-op day 3 and day 5 respectively. The test will be performed twice on post-op day 3 and post-op day 5 with 6 hours minimum gap in between to promote patient recovery and test re-test reliability. Participants pre-test and post-test vitals will be taken and their test outcomes readings will be noted on the self-administered questionnaire.
  Interventions: Other: Physiotherapy Protocol

INTERVENTIONS:
Other: Physiotherapy Protocol — Each participant consenting to the study will be given a physiotherapy session on post-op day 1 and day 2 by a physiotherapist. The session will include bed mobility exercises including active ROM exercises of all extremities, breathing exercises, nebulization and chest physical therapy, incentive spirometer. Progressing to supported sitting at the edge of bed, sitting on a chair under supervision, supported walk inside the room , sitting independently in chair and lastly before discharge climbing 2 flights of stair.

SUMMARY:
The purpose of this research is to determine which performance based functional outcome test among Time up and go test, Five times sit to stand test, 2 minute walk test and 6 minute walk test has the greatest significance in improving functional outcomes in post-CABG surgery patients.

DETAILED DESCRIPTION:
Coronary artery disease is the leading cause of death worldwide and has adverse effects on functionality. It causes functional limitations which affects the cardiac output resulting in reduced morbidity and mortality. To improve the life expectancy, an invasive surgical procedure is done known as CABG. To reduce the chances of reoccurrence of coronary artery disease post- CABG surgery patients are enrolled in the Cardiac Rehab program which focuses on improving quality of life of the patient, to increase life expectancy, improve functional independence and reduce chances of graft failure. In Cardiac Rehabilitation our focus would be on identifying the performance based functional outcome measure test which demonstrates the greatest clinimetric significance in improving functional outcome measure in post- CABG patients. The four clinimetric tests used in this research are time up and go test, five times sit to stand test, 2 minute walk test and 6 minute walk test on post operative day 3 and day 5 respectively. The result of this research would indicate which test is most significant in enhancing functionality of post-CABG patients providing valuable and evidence-based approach for healthcare providers to design rehabilitation protocols.

ELIGIBILITY:
Inclusion Criteria:

* 30-50 years old
* Post-op CABG patients
* Include male and female both
* Mobile patients
* Post-op day 3 and day 5 of CABG surgery

Exclusion Criteria:

* Occurrence of adverse events
* Unstable hemodynamically
* Patients with documented cognitive dysfunction
* Patients with neurologic or musculoskeletal disease (excluding osteoarthritis) that adversely affects gait or weight-bearing
* Patients with severe co-morbidities, recurrent attacks, and unstable condition.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Time up and go test | 6 hours
  On post op- day 3 and 5 Participants will quickly perform test to assess lower extremity strength and risk of fall. The time taken to complete test will be noted
Five times sit to stand test | 6 hours
  On post-op day 3 and 5, Participants will perform test by transitioning from sitting to standing five times in row, time would be noted. This test helps to evaluate lower extremity balance and strength.
2 Minute walk test | 6 hours
  The test will be performed on post-op day 3 and 5, the participants will walk on a flat surface in a straight line and the distance will be noted. This test assess endurance
6 Minute walk test | 6 hours
  This is a self-paced test which will be performed on post-op day 3 and 5 where the participants have walk on a flat, smooth surface. The distance covered during this test will be noted. It measures aerobic capacity and endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD, Principal Investigator — Riphah International University
Locations (1):
- Armed Forces Institute of Cardiology, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melo TA, Duarte ACM, Bezerra TS, Franca F, Soares NS, Brito D. The Five Times Sit-to-Stand Test: safety and reliability with older intensive care unit patients at discharge. Rev Bras Ter Intensiva. 2019;31(1):27-33. doi: 10.5935/0103-507X.20190006. Epub 2019 Mar 14. PMID 30892478
- [Background] Rodrigues F, Teixeira JE, Forte P. The Reliability of the Timed Up and Go Test among Portuguese Elderly. Healthcare (Basel). 2023 Mar 23;11(7):928. doi: 10.3390/healthcare11070928. PMID 37046858
- [Background] de Jesus SFC, Bassi-Dibai D, Pontes-Silva A, da Silva de Araujo A, de Freitas Faria Silva S, Veneroso CE, de Paula Gomes CAF, Dibai-Filho AV. Construct validity and reliability of the 2-Minute Step Test (2MST) in individuals with low back pain. BMC Musculoskelet Disord. 2022 Dec 5;23(1):1062. doi: 10.1186/s12891-022-06050-w. PMID 36471309
- [Background] Giannitsi S, Bougiakli M, Bechlioulis A, Kotsia A, Michalis LK, Naka KK. 6-minute walking test: a useful tool in the management of heart failure patients. Ther Adv Cardiovasc Dis. 2019 Jan-Dec;13:1753944719870084. doi: 10.1177/1753944719870084. PMID 31441375
- [Background] Essop-Adam A, Daynes E, Houghton JSM, Nickinson ATO, Sayers RDS, Haunton VJ, Pepper C, Singh SJ. Clinimetrics of performance-based functional outcome measures for vascular amputees: A systematic review. Ann Phys Rehabil Med. 2023 Sep;66(6):101756. doi: 10.1016/j.rehab.2023.101756. Epub 2023 Jun 3. PMID 37276748
- [Background] Osailan A, Abdelbasset WK. Exercise-based cardiac rehabilitation for postcoronary artery bypass grafting and its effect on hemodynamic responses and functional capacity evaluated using the Incremental Shuttle Walking Test: A retrospective pilot analysis. J Saudi Heart Assoc. 2020 Apr 17;32(1):25-33. doi: 10.37616/2212-5043.1005. eCollection 2020. PMID 33154888
- [Background] Puri SN, Lalwani L. A Comparison Between Cardiac Telerehabilitation Program and Outpatient Hospital-Based Cardiac Rehabilitation Program for Patients Undergoing Coronary Artery Bypass Graft (CABG) Surgery: A Review. Cureus. 2023 Nov 8;15(11):e48488. doi: 10.7759/cureus.48488. eCollection 2023 Nov. PMID 38073989